CLINICAL TRIAL: NCT04627324
Title: Efficacy of Using 3D Motion Tracking Toothbrush in Dental Plaque Control
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yonsei University (Other)
Collaborators: National Research Foundation of Korea (Other)
Responsible Party: Principal Investigator, Kee-Deog Kim, Professor, Yonsei University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2-2008-0005
Record Dates: First submitted 2020-11-02; First posted 2020-11-13 (Actual); Last update posted 2020-11-17 (Actual); Status verified 2020-11

CONDITIONS: Toothbrushing
Keywords: Teledentistry; Schoolchildren; Oral hygiene; Computer; Smart toothbrush; Dental plaque
MeSH Terms: conditions — Dental Plaque | interventions — Microscopy, Scanning Tunneling; Drug Delivery Systems

STUDY DESIGN:
Who Masked: Investigator
Masking Description: A dental hygienist blinded to group assignment determined plaque status. Participants were randomly assigned into two equally sized groups by flipping a coin.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The smart toothbrush and smart mirror (STM) system toothbrushing instruction (TBI) (Experimental): Participants received using the STM system TBI. The plaque indexes were evaluated at baseline, immediately after TBI (day 0), 1 week, 1 month and 10 month (1st study only) after TBI.
  Interventions: Device: The smart toothbrush and smart mirror (STM) system (XiuSolution, Gyeonggi-do, Korea)
- conventional toothbrushing instruction (TBI) (Active Comparator): Participants received using conventional TBI. The plaque indexes were evaluated at baseline, immediately after TBI (day 0), 1 week, 1 month and 10 month (1st study only) after TBI.
  Interventions: Device: Conventional toothbrush

INTERVENTIONS:
Device: The smart toothbrush and smart mirror (STM) system (XiuSolution, Gyeonggi-do, Korea) — The STM system comprises a smart mirror, which is integrated into a computer monitor, and a 3D motion-capture device inside of a modified toothbrush holder. The computer program displays a toothbrushing animation in the mirror. Toothbrush motions detected by sensors embedded inside the holder are captured and sent to the server for analysis.
  (used only during the test visits)
  Participants had to brush their teeth at home (using toothbrushes with a flat-trimmed nylon bristle of identical type and length.) for 3 min thrice daily, after meals, as recommended by the Korean Dental Association.
  Arms: The smart toothbrush and smart mirror (STM) system toothbrushing instruction (TBI)
Device: Conventional toothbrush — toothbrushes with a flat-trimmed nylon bristle of identical type and length.
  Participants had to brush their teeth at home for 3 min thrice daily, after meals, as recommended by the Korean Dental Association.
  Arms: conventional toothbrushing instruction (TBI)

SUMMARY:
The objective of this study was to compare the efficacy of computer-assisted TBI (toothbrushing instruction) using a smart toothbrush and smart mirror (STM system) in plaque control to that of conventional TBI.

DETAILED DESCRIPTION:
The STM system comprises a smart mirror, which is integrated into a computer monitor, and a 3D motion-capture device inside of a modified toothbrush holder. The computer program displays a toothbrushing animation in the mirror. Toothbrush motions detected by sensors embedded inside the holder are captured and sent to the server for analysis.

The investigators evaluated the efficacy of TBI with a STM system by analyzing the reductions of the modified Quigley-Hein plaque index in

1. st study - 60 volunteers (adults) - The data for which have been published (reference)
2. nd study - 42 volunteers (schoolchildren) - manuscript prepared
3. rd study - 60 volunteers (adults and children)

These participants were separated randomly into two groups: conventional TBI (control group) and STM system TBI (experimental group).

The changes in the plaque indexes were recorded immediately, 1 week, 1 month, and 10 months (1st study only) after TBI.

ELIGIBILITY:
Inclusion Criteria:

* Participants with poor oral conditions need more toothbrush instruction
* Participants were required to have their gingivitis and baseline plaque scores >1.5 (the Turesky Modification of the Quigley-Hein index)

Exclusion Criteria:

* if they had gross dental caries or orthodontic appliances, or were medically compromised.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 209 (Actual)
Dates: Start 2008-09-01 (Actual); Primary Completion 2011-08-01 (Actual); Study Completion 2011-08-01 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in plaque index at 10 month after TBI (1st study-adults) | Baseline, immediately after TBI (day 0), 1 week, 1 month and 10 month after TBI.
  The effects of smart toothbrush and smart mirror (STM) system TBI and conventional TBI on dental plaque in adults were compared in this study.
  Plaque examination was scored on the buccal and lingual surface of all teeth. The Turesky Modification of the Quigley-Hein index was scored between 0 (no plaque) and 5 (plaque covering ≥ two-thirds of the tooth crown) The percentages of plaque removal at each surfaces and whole mouth were determined with the formula: percentage plaque reduction = pre-post / pre X100 (pre=prebrushing plaque value; post=postbrushing plaque value).
Change from Baseline in plaque index at 1 month after TBI (2nd study-schoolchildren) | Baseline, immediately after TBI (day 0), 1 week, 1 month after TBI.
  The effects of smart toothbrush and smart mirror (STM) system TBI and conventional TBI on dental plaque in schoolchildren were compared in this study.
  Plaque examination was scored on the buccal and lingual surface of all teeth (if a permanent tooth had not erupted yet, the primary tooth in the corresponding area was tested).
  The Turesky Modification of the Quigley-Hein index was scored between 0 (no plaque) and 5 (plaque covering ≥ two-thirds of the tooth crown) The percentages of plaque removal at each surfaces and whole mouth were determined with the formula: percentage plaque reduction = pre-post / pre X100 (pre=prebrushing plaque value; post=postbrushing plaque value).
Change from Baseline in plaque index at 1 month after TBI (3rd study-adults and children) | Baseline, immediately after TBI (day 0), 1 week, 1 month after TBI.
  The effects of smart toothbrush and smart mirror (STM) system TBI and conventional TBI on dental plaque in adults and children were compared in this study.
  Plaque examination was scored on the buccal and lingual surface of all teeth (if a permanent tooth had not erupted yet, the primary tooth in the corresponding area was tested).
  The Turesky Modification of the Quigley-Hein index was scored between 0 (no plaque) and 5 (plaque covering ≥ two-thirds of the tooth crown) The percentages of plaque removal at each surfaces and whole mouth were determined with the formula: percentage plaque reduction = pre-post / pre X100 (pre=prebrushing plaque value; post=postbrushing plaque value).

CONTACTS AND LOCATIONS:
Overall Officials: Kee-Deog Kim, PhD, Study Chair — Department of Advanced General Dentistry College of Dentistry, Yonsei University, Seoul, Korea

REFERENCES:
- [Result] Kim KD, Jeong JS, Lee HN, Gu Y, Kim KS, Lee JW, Park W. Efficacy of computer-assisted, 3D motion-capture toothbrushing instruction. Clin Oral Investig. 2015 Jul;19(6):1389-94. doi: 10.1007/s00784-014-1350-y. Epub 2014 Nov 14. PMID 25391495
- [Derived] Jeong JS, Kim KS, Lee JW, Kim KD, Park W. Efficacy of tooth brushing via a three-dimensional motion tracking system for dental plaque control in school children: a randomized controlled clinical trial. BMC Oral Health. 2022 Dec 22;22(1):626. doi: 10.1186/s12903-022-02665-6. PMID 36550451